CLINICAL TRIAL: NCT00922623
Title: A Multicenter Study of The Safety and Effectiveness of Dermal Filler, Belotero®, After Mid-to-Deep Dermal Implantation for Correction of Moderate to Severe Facial Wrinkles (Such as Nasolabial Folds) Over 24 Weeks in Subjects With Fitzpatrick Phototype Scores of IV, V, and VI.
Brief Title: Safety and Effectiveness of Belotero® in Subjects With Fitzpatrick Phototypes IV Through VI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Merz North America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MUS 90028-0622/1 Supplement
Record Dates: First submitted 2009-06-03; First posted 2009-06-17 (Estimated); Results first posted 2012-01-30 (Estimated); Last update posted 2013-04-26 (Estimated); Status verified 2013-04

CONDITIONS: Facial Wrinkles
Keywords: Nasolabial folds

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Belotero® (Experimental)
  Interventions: Device: Belotero®

INTERVENTIONS:
Device: Belotero® — Hyaluronic acid dermal filler, Belotero®, single use syringe, injected into mid to deep dermal layer
  Other Names: Nasolabial folds

SUMMARY:
This is a study to assess how safe and effective an investigational product, Belotero® is in people with all skin types with facial wrinkles, such as nasolabial folds. Nasolabial folds are wrinkles on the face that go from outside of the nostrils to the edges of the mouth.

DETAILED DESCRIPTION:
The Fitzpatrick Skin Phototype Scale goes from number 1 (I), which is the very lightest skin tone, to number 6 (VI) which is the very darkest skin tone. This study is to determine the safety and effectiveness of Belotero® in people with skin phototypes of 1(I)thru 6 (VI).

ELIGIBILITY:
Inclusion Criteria:

1. Had reviewed and signed a statement of Informed Consent and HIPAA authorization. In addition, subjects were asked to provide a separate release for use of their photographs in publications. Subjects had a right to refuse the photo release without jeopardizing their eligibility to participate in the study.
2. Was 18 to 75 years of age, of any race or sex.
3. If female, was post-menopausal for at least one year; or had undergone a hysterectomy; or a tubal ligation; or if of childbearing potential, had negative urine pregnancy test results and agreed to use an approved method of birth control throughout the study (ie, oral/systemic contraceptives, intrauterine device [IUD], or spermicide in combination with a barrier method of contraception), or was abstinent, or was in a monogamous relationship with a partner who had had a vasectomy.
4. Had bilateral nasolabial folds with a severity of 2 or 3 on the wrinkle severity rating scale (SRS) as assessed by the Evaluator Investigator.
5. Subjects were to have been rated IV, V, or VI on the Fitzpatrick Skin Phototype Scale.
6. Had adequate understanding of the language (spoken and written English or Spanish) and was willing to comply with the study requirements.

Exclusion Criteria:

1. A personal history of allergic/anaphylactic reactions including hypersensitivity to local anesthetics (eg, lidocaine, etc), hyaluronic acid (HA) preparations, and/or gram-positive bacterial protein.
2. A known history of keloids or bleeding disorders.
3. Leukoderma (vitiligo) or a family history of leukoderma or other pigmentary disorders.
4. An active inflammatory process in the nasolabial fold area (skin eruptions such as cysts, pimples, rashes, cancerous/pre-cancerous lesions, psoriasis, neurodermatitis, or any other active skin disease) or severe scarring that might interfere with study assessments.
5. If female, pregnant, planning to become pregnant during the study, or breast feeding.
6. Planned to undergo major facial surgery during the course of the study (eg, rhinoplasty [with or without implant], facelift, congenital defect repair, etc).
7. Clinically important disease, as judged by the investigator, within 3 months of the study (eg, significant laboratory test abnormalities, myocardial infarct, stroke, cancer, connective tissue diseases [scleroderma, systemic lupus erythematous], systemic infection, uncontrolled diabetes, etc.), including those with medical conditions that might require the use of immunosuppressive medications during the trial (eg, severe, uncontrolled asthma, rheumatoid arthritis, autoimmune diseases, etc).
8. Severe physical, neurological or mental disease.
9. Excessive facial hair that might interfere with the evaluation of the wrinkle assessments.
10. Any systemic or dermatologic disorder, which, in the opinion of the investigator, would interfere with the study results or increase the risk of AEs.
11. Had used exclusionary medications/treatments.
12. Participation in a clinical investigation within the 30 days prior to the first planned device administration or during this trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2009-05; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rhoda Narins, MD, Principal Investigator — Dermatology Surgery and Laser Center
Locations (3):
- United States (3):
  - Pearl E Grimes, Los Angeles, California
  - Valerie Callender, Mitchellville, Maryland
  - Jeanine B Downie, Montclair, New Jersey

RESULTS

PARTICIPANT FLOW:
Groups:
- Belotero®: Belotero® injection into both nasolabial folds of Fitzpatrick IV, V, VI subjects.
Period: Overall Study
Arm/Group | Belotero®
Started | 93
Completed | 88
Not Completed | 5
Not completed — Other | 4
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Belotero®
Number analyzed (Participants) | 93
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 81
  >=65 years | 12
Age Continuous [Mean (Standard Deviation); unit: years] | 51.5 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80
  Male | 13
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 90
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Product-related Adverse Events.
Description: Adverse events considered possibly, probably, or definitely related to study product are summarized by body system and MedDRA preferred term.
Time Frame: 24 weeks
Population: The Full Analysis Set (FAS) consisted of all subjects enrolled and treated with Belotero (ITT principle).
Measure: Number; unit: percentage of subjects with AEs.
Groups:
- Belotero, Left Nasolabial Fold: Belotero injected into the Left Nasolabial Fold of the Face
- Belotero, Right Nasolabial Fold: Belotero injected into the Right Nasolabial Fold of the Face
Arm/Group | Belotero, Left Nasolabial Fold | Belotero, Right Nasolabial Fold
Number analyzed (Participants) | 93 | 93
percentage of subjects with AEs. | 71 | 72

ADVERSE EVENTS:
Arm/Group | Belotero, Left Nasolabial Fold | Belotero, Right Nasolabial Fold
Serious Adverse Events (participants affected / at risk) | 0/93 | 0/93
Other Adverse Events (participants affected / at risk) | 71/93 | 72/93
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Belotero, Left Nasolabial Fold (N=93) | Belotero, Right Nasolabial Fold (N=93)
Injection site swelling (General disorders) | 55 | 56
Injection site induration (General disorders) | 51 | 55
Injection site pain (General disorders) | 37 | 47
Injection site nodule (General disorders) | 31 | 38
Injection site erythema (General disorders) | 29 | 29
Injection site pruritus (General disorders) | 19 | 22
Injection site bruising (General disorders) | 14 | 22
Injection site discoloration (General disorders) | 15 | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any proposed press release, announcement, disclosure for publication, whether or not in writing, prepared by or on behalf of Consultant as part of services under this Agreement or that relates to the work performed hereunder must be reviewed and approved in writing by Merz prior to dissemination.